CLINICAL TRIAL: NCT00038948
Title: A Randomized, Open-label, Comparative Evaluation of Conversion From Calcineurin Inhibitors to Sirolimus Versus Continued Use of Calcineurin Inhibitors in Renal Allograft Recipients
Brief Title: Study Comparing Conversion to Sirolimus vs. Continued Use of Calcineurin Inhibitors in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-316
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-04

CONDITIONS: Renal Transplantation
Keywords: Renal; Allograft; Recipients
MeSH Terms: interventions — Sirolimus; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Conversion from calcineurin inhibitor immunosuppression to Sirolimus-based immunosuppression
  Interventions: Drug: Sirolimus; Drug: tacrolimus; Drug: Cyclosporine A
- B (Active Comparator): Continued calcineurin inhibitor therapy
  Interventions: Drug: Sirolimus; Drug: tacrolimus; Drug: Cyclosporine A

INTERVENTIONS:
Drug: Sirolimus — Sirolimus, Cyclosporine A & Tacrolimus are concentration controlled
Drug: tacrolimus
Drug: Cyclosporine A

SUMMARY:
The purpose of this study is to determine the effect of conversion from calcineurin inhibitor to sirolimus based therapy on renal function.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 13 years.
* Receiving CsA or tacrolimus from the time of transplantation or within 2 weeks thereafter
* Patients with a functioning allograft and a Nankivell GFR greater than or equal to 20 mL/min, within 2 weeks before randomization

Exclusion Criteria:

* Biopsy-confirmed acute rejection within 12 weeks before randomization, that was determined to require antirejection treatment
* Patients in whom kidney-pancreas or other multiple organ transplants have been performed

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2002-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Reichen J, Stickel F, Bhattacharya I, Matschke K, Maller E, Korth-Bradley J. Repeat-dose sirolimus pharmacokinetics and pharmacodynamics in patients with hepatic allografts. Eur J Clin Pharmacol. 2012 May;68(5):589-97. doi: 10.1007/s00228-011-1172-7. Epub 2011 Dec 6. PMID 22143911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from January 2002 to September 2003.
Pre-assignment Details: Patients were screened for two weeks.
Groups:
- SRL Conversion in Stable Renal Transplant Recipients: Conversion from calcineurin inhibitor immunosuppression therapy to Sirolimus-based immunosuppression therapy.
- CNI Continuation in Stable Renal Transplant Recipients: Continued calcineurin inhibitor immunosuppression therapy
Period: Overall Study
Arm/Group | SRL Conversion in Stable Renal Transplant Recipients | CNI Continuation in Stable Renal Transplant Recipients
Started | 555 | 275
Completed | 386 | 198
Not Completed | 169 | 77
Not completed — Adverse Event | 131 | 43
Not completed — Lost to Follow-up | 4 | 4
Not completed — Nonmedical event | 5 | 7
Not completed — Withdrawal by Subject | 23 | 10
Not completed — Protocol Violation | 3 | 7
Not completed — Lack of Efficacy | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRL Conversion in Stable Renal Transplant Recipients | CNI Continuation in Stable Renal Transplant Recipients | Total
Number analyzed (Participants) | 555 | 275 | 830
Age Continuous [Median (Full Range); unit: years] | 45.00 [13.20 to 75.10] | 43.50 [12.80 to 74.00] | 44.50 [12.80 to 75.10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 81 | 251.0
  Male | 385 | 194 | 579.0

OUTCOME MEASURES:

1. Primary Outcome: Nankivell Glomerular Filtration Rate (GFR)
Description: Nankivell GFR: patients with baseline GFR of 20.0 to 40.0 mL/min and patients with baseline GFR of greater than 40.0 mL/min. GFR is an index of kidney function. A higher value means better kidney function.
Time Frame: 52 weeks
Population: Patients were stratified by GFR at baseline. GFR 20-40 mL/min and GFR >40 mL/min.
Measure: Mean (Standard Error); unit: mL/min
Groups:
- SRL Conversion Strata 20.0-40.0 mL/Min: Conversion from calcineurin inhibitor immunosuppression therapy to Sirolimus-based immunosuppression therapy in stable renal transplant recipients
- CNI Continuation Strata 20.0-40.0 mL/Min; CNI Continuation Strata >40.0 mL/Min: Continued calcineurin inhibitor immunosuppression therapy in renal transplant recipients.
- SRL Conversion Strata >40.0 mL/Min: Conversion from calcineurin inhibitor immunosuppression therapy to Sirolimus-based immunosuppression therapy in renal transplant recipients.
Arm/Group | SRL Conversion Strata 20.0-40.0 mL/Min | CNI Continuation Strata 20.0-40.0 mL/Min | SRL Conversion Strata >40.0 mL/Min | CNI Continuation Strata >40.0 mL/Min
Number analyzed (Participants) | 58 | 29 | 496 | 245
mL/min | 24.56 (2.42) | 27.24 (3.71) | 59.04 (0.89) | 57.73 (1.1)
Statistical Analysis 1: Comparison: SRL Conversion Strata 20.0-40.0 mL/Min vs CNI Continuation Strata 20.0-40.0 mL/Min; Baseline GFR of 20.0 to 40.0 mL/min; Test type: Superiority or Other; p = 0.575, ANCOVA — Analysis of covariance p-value; Weighted difference = -2.68, 95% CI [-12.27 to 6.91] — Data was adjusted for baseline and center
Statistical Analysis 2: Comparison: SRL Conversion Strata >40.0 mL/Min vs CNI Continuation Strata >40.0 mL/Min; Baseline GFR of >40.0 mL/min; Test type: Superiority or Other; p = 0.278, ANCOVA — Analysis of covariance p-value; Weighted difference = 1.31, 95% CI [-1.06 to 3.69] — Data was adjusted for baseline and center

2. Secondary Outcome: First Occurrence of Biopsy-confirmed Acute Rejection, Graft Loss, or Death.
Description: Number of patients who experienced for the first time either biopsy-confirmed acute rejection, graft loss, or death by weeks 52 and 104. Assessed by individual endpoint and as composite endpoint (all combined).
Time Frame: 52 and 104 weeks
Population: Patients were stratified by GFR at baseline. GFR 20-40 mL/min and GFR >40 mL/min.
Measure: Number; unit: patients
Groups:
- SRL Conversion Strata 20.0-40.0 mL/Min; SRL Conversion Strata >40.0 mL/Min: Conversion from calcineurin inhibitor immunosuppression to Sirolimus-based immunosuppression
- CNI Continuation Strata 20.0-40.0 mL/Min; CNI Continuation Strata >40.0 mL/Min: Continued calcineurin inhibitor therapy
Arm/Group | SRL Conversion Strata 20.0-40.0 mL/Min | CNI Continuation Strata 20.0-40.0 mL/Min | SRL Conversion Strata >40.0 mL/Min | CNI Continuation Strata >40.0 mL/Min
Number analyzed (Participants) | 58 | 29 | 497 | 246
patients
  52 weeks - Acute rejection | 4 | 0 | 8 | 3
  52 weeks - Graft loss | 7 | 3 | 3 | 3
  52 weeks - Death | 3 | 0 | 6 | 1
  52 weeks - Missing | 0 | 0 | 5 | 1
  104 weeks - Acute rejection | 5 | 1 | 27 | 9
  104 weeks - Graft loss | 12 | 9 | 12 | 8
  104 weeks - Death | 7 | 0 | 13 | 3
  104 weeks - Missing | 0 | 2 | 13 | 8
Statistical Analysis 1: Comparison: SRL Conversion Strata 20.0-40.0 mL/Min vs CNI Continuation Strata 20.0-40.0 mL/Min vs SRL Conversion Strata >40.0 mL/Min vs CNI Continuation Strata >40.0 mL/Min; 52 weeks statistical analysis across strata; Test type: Superiority or Other; p = 0.135, Cochran-Mantel-Haenszel — Tests the equality of rates between treatments across strata at 52 weeks
Statistical Analysis 2: Comparison: SRL Conversion Strata 20.0-40.0 mL/Min vs CNI Continuation Strata 20.0-40.0 mL/Min vs SRL Conversion Strata >40.0 mL/Min vs CNI Continuation Strata >40.0 mL/Min; 104 weeks statistical analysis across strata; Test type: Superiority or Other; p = 0.559, Cochran-Mantel-Haenszel — Tests the equality of rates between treatments across strata at 104 weeks

ADVERSE EVENTS:
Arm/Group | SRL Conversion in Stable Renal Transplant Recipients | CNI Continuation in Stable Renal Transplant Recipients
Serious Adverse Events (participants affected / at risk) | 81/551 | 45/273
Other Adverse Events (participants affected / at risk) | 545/551 | 264/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRL Conversion in Stable Renal Transplant Recipients (N=551) | CNI Continuation in Stable Renal Transplant Recipients (N=273)
Abdominal pain (General disorders) | 19 | 5
Abdominal syndrome acute (General disorders) | 3 | 2
Abscess (General disorders) | 7 | 2
Accidental injury (General disorders) | 14 | 3
Accidental overdose (General disorders) | 2 | 1
Allergic reaction (General disorders) | 1 | 0
Ascites (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Back pain (General disorders) | 2 | 2
Carcinoma (General disorders) | 0 | 1
Cellulitis (General disorders) | 10 | 3
Chest pain (General disorders) | 8 | 2
Chills (General disorders) | 5 | 0
Chills and fever (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Drug level increased (General disorders) | 1 | 0
Face edema (General disorders) | 2 | 0
Fever (General disorders) | 43 | 10
Flu syndrome (General disorders) | 4 | 0
Gangrene (General disorders) | 2 | 0
Generalized edema (General disorders) | 3 | 0
Granuloma (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Hernia (General disorders) | 5 | 2
Infection (General disorders) | 40 | 8
Lab test abnormal (General disorders) | 3 | 0
Lymphocele (General disorders) | 1 | 0
Moniliasis (General disorders) | 1 | 0
Neck pain (General disorders) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Overdose (General disorders) | 4 | 1
Pain (General disorders) | 2 | 1
Pelvic pain (General disorders) | 0 | 1
Peritonitis (General disorders) | 2 | 1
Sepsis (General disorders) | 17 | 5
Septic shock (General disorders) | 3 | 1
Suicide attempt (General disorders) | 1 | 0
Transplant rejection (General disorders) | 18 | 4
Aneurysm (Cardiac disorders) | 2 | 3
Angina pectoris (Cardiac disorders) | 2 | 1
Aortic stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arterial anomaly (Vascular disorders) | 4 | 1
Arteriosclerosis (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 3 | 0
Cardiovascular disorder (Cardiac disorders) | 2 | 2
Cerebral ischemia (Vascular disorders) | 0 | 2
Cerebrovascular accident (Vascular disorders) | 5 | 3
Congestive heart failure (Cardiac disorders) | 6 | 2
Coronary artery disorder (Cardiac disorders) | 3 | 1
Cyanosis (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 8 | 3
Embolus (Vascular disorders) | 1 | 1
Endocarditis (Cardiac disorders) | 1 | 0
Heart arrest (Cardiac disorders) | 6 | 2
Heart failure (Cardiac disorders) | 5 | 1
Hemorrhage (Vascular disorders) | 2 | 1
Hypertension (Cardiac disorders) | 13 | 4
Hypervolemia (Vascular disorders) | 5 | 1
Hypotension (Cardiac disorders) | 1 | 3
Hypovolemia (Vascular disorders) | 3 | 1
Infarct (Cardiac disorders) | 0 | 1
Migraine (Cardiac disorders) | 1 | 0
Myocardial infarct (Cardiac disorders) | 2 | 0
Occlusion (Vascular disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 2
Peripherial gangrene (Vascular disorders) | 2 | 1
Peripherial vascual disorder (Vascular disorders) | 6 | 4
Phlebitis (Vascular disorders) | 1 | 0
Pulmonary embolus (Cardiac disorders) | 3 | 1
Shock (Cardiac disorders) | 4 | 0
Subarachnoid hemorrhage (Vascular disorders) | 2 | 0
Syncope (Cardiac disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 4 | 3
Thrombosis (Vascular disorders) | 2 | 3
Valvular heart disease (Cardiac disorders) | 1 | 0
Vascular disorder (Vascular disorders) | 2 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 0
Bloody diarrhea (Gastrointestinal disorders) | 1 | 0
Carcinoma of the mouth (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholelithiasis (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 8 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 36 | 3
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitits (Gastrointestinal disorders) | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 5 | 0
Gastroenteritis (Gastrointestinal disorders) | 28 | 4
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal disorder general (Gastrointestinal disorders) | 3 | 2
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 | 1
Hematemesis (Gastrointestinal disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal nercosis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Liver damage (Hepatobiliary disorders) | 1 | 0
Liver function tests abnormal (Hepatobiliary disorders) | 8 | 0
Liver tenderness (Hepatobiliary disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
Mouth ulcerations (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 1
Nausea and vomiting (Gastrointestinal disorders) | 0 | 2
Oral moniliasis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Hepatobiliary disorders) | 2 | 1
Rectal disorder (Gastrointestinal disorders) | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Ulcerative colitis (Gastrointestinal disorders) | 1 | 0
Ulcerative proctitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 3
Parathyroid disorder (Metabolism and nutrition disorders) | 4 | 3
Anemia (Blood and lymphatic system disorders) | 21 | 3
Aplastic anemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0
International normalized ratio increased (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 0
Luekocytosis (Blood and lymphatic system disorders) | 1 | 0
Luekopenia (Blood and lymphatic system disorders) | 4 | 0
Lymphadenopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma like reaction (Blood and lymphatic system disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Blood uria nitrogren increased (Metabolism and nutrition disorders) | 9 | 3
Acidosis (Metabolism and nutrition disorders) | 2 | 0
Amyloidosis (Metabolism and nutrition disorders) | 1 | 0
Calcium disorder (Metabolism and nutrition disorders) | 1 | 0
Creatinine increased (Metabolism and nutrition disorders) | 36 | 9
Dehydration (Metabolism and nutrition disorders) | 14 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 2
Edema (Metabolism and nutrition disorders) | 3 | 0
Electrolyte abnormality (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Healing abnormal (Metabolism and nutrition disorders) | 5 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypercholesteremia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Peripheral edema (Metabolism and nutrition disorders) | 9 | 2
Respiratory acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone necrosis (Musculoskeletal and connective tissue disorders) | 6 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Myasthenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Necrotising faciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Central nervous system anomaly (Nervous system disorders) | 0 | 1
Agitation (Nervous system disorders) | 1 | 0
Confusion (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 1 | 2
Depression (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hostility (Nervous system disorders) | 1 | 0
Meningitis (Nervous system disorders) | 2 | 0
Nerve root compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0
Neuropathy (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Vocal chord paralysis (Nervous system disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive airway disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough increased (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Lung edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Mediastinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Pluritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 57 | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder general (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Fungal dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Herpes simplex (Skin and subcutaneous tissue disorders) | 5 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 6 | 2
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Skin benign neoplasm (Skin and subcutaneous tissue disorders) | 0 | 1
Skin carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 15
Skin disorder general (Skin and subcutaneous tissue disorders) | 2 | 2
Skin granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 1
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract specified (Eye disorders) | 1 | 0
Otitis externa (Ear and labyrinth disorders) | 1 | 0
Otitis media (Ear and labyrinth disorders) | 3 | 0
Parosmia (Eye disorders) | 1 | 0
Acute kidney failure (Renal and urinary disorders) | 11 | 4
Albuminuria (Renal and urinary disorders) | 8 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Glomerulitis (Renal and urinary disorders) | 5 | 2
Hematuria (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 6 | 0
Hydroureter (Renal and urinary disorders) | 0 | 1
Kidney calculus (Renal and urinary disorders) | 1 | 0
Kidney failure (Renal and urinary disorders) | 13 | 9
Kidney function abnormal (Renal and urinary disorders) | 29 | 18
Kidney tubular disorder (Renal and urinary disorders) | 1 | 0
Kidney tubular necrosis (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 3 | 1
Metrorrhagia (Renal and urinary disorders) | 3 | 1
Nephritis (Renal and urinary disorders) | 3 | 1
Nephrosclerosis (Renal and urinary disorders) | 3 | 0
Nephrosis (Renal and urinary disorders) | 9 | 0
Oliguria (Renal and urinary disorders) | 2 | 0
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Polycystic kidney (Renal and urinary disorders) | 1 | 0
Prostatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Pyelonephritis (Renal and urinary disorders) | 12 | 4
Scrotal edema (Renal and urinary disorders) | 1 | 0
Toxic nephropathy (Renal and urinary disorders) | 1 | 0
Unintended pregnancy (Reproductive system and breast disorders) | 1 | 1
Uremia (Renal and urinary disorders) | 4 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 2 | 1
Urinary tract infection (Renal and urinary disorders) | 33 | 12
Local reaction to procedure (Injury, poisoning and procedural complications) | 16 | 7
Device malfunction (General disorders) | 3 | 0
Other etiology unknown (General disorders) | 0 | 2
Cholecystitis (Gastrointestinal disorders) | 1 | 0
Pancreas disorder (Hepatobiliary disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | SRL Conversion in Stable Renal Transplant Recipients (N=551) | CNI Continuation in Stable Renal Transplant Recipients (N=273)
Abdominal pain (General disorders) | 87 | 42
Accidental injury (General disorders) | 98 | 39
Asthenia (General disorders) | 75 | 30
Back pain (General disorders) | 46 | 37
Chest pain (General disorders) | 42 | 23
Cyst (General disorders) | 30 | 13
Face edema (General disorders) | 32 | 2
Fever (General disorders) | 125 | 28
Flu syndrome (General disorders) | 25 | 14
Headache (General disorders) | 111 | 43
Lab test abnormal (General disorders) | 38 | 15
Pain (General disorders) | 82 | 38
Transplant rejection (General disorders) | 32 | 14
Hypertension (Cardiac disorders) | 127 | 68
Anorexia (Gastrointestinal disorders) | 33 | 11
Aphthous stomatitis (Gastrointestinal disorders) | 49 | 3
Constipation (Gastrointestinal disorders) | 32 | 15
Diarrhea (Gastrointestinal disorders) | 234 | 75
Dyspepsia (Gastrointestinal disorders) | 35 | 21
Gastritis (Gastrointestinal disorders) | 21 | 14
Gum hyperplasia (Gastrointestinal disorders) | 1 | 15
Liver function tests abnormal (Gastrointestinal disorders) | 38 | 4
Mouth ulceration (Gastrointestinal disorders) | 34 | 1
Nausea (Gastrointestinal disorders) | 69 | 27
Stomatitis (Gastrointestinal disorders) | 59 | 3
Vomiting (Gastrointestinal disorders) | 72 | 38
Diabetes mellitus (Endocrine disorders) | 33 | 12
Anemia (Blood and lymphatic system disorders) | 219 | 61
Ecchymosis (Blood and lymphatic system disorders) | 28 | 5
Iron deficiency anemia (Blood and lymphatic system disorders) | 32 | 3
Leukopenia (Blood and lymphatic system disorders) | 75 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 79 | 10
Acidosis (Metabolism and nutrition disorders) | 28 | 15
BUN increased (Metabolism and nutrition disorders) | 34 | 13
Creatinine increased (Metabolism and nutrition disorders) | 113 | 48
Dehydration (Metabolism and nutrition disorders) | 35 | 6
Edema (Metabolism and nutrition disorders) | 62 | 18
Gout (Metabolism and nutrition disorders) | 29 | 15
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 15
Hypercholesteremia (Metabolism and nutrition disorders) | 245 | 44
Hyperglycemia (Metabolism and nutrition disorders) | 76 | 20
Hyperkalemia (Metabolism and nutrition disorders) | 13 | 19
Hyperlipemia (Metabolism and nutrition disorders) | 317 | 83
Hyperuricemia (Metabolism and nutrition disorders) | 46 | 48
Hypokalemia (Metabolism and nutrition disorders) | 57 | 8
Lactic dehydrogenase increased (Metabolism and nutrition disorders) | 70 | 6
Peripheral edema (Metabolism and nutrition disorders) | 190 | 51
SGOT increased (Metabolism and nutrition disorders) | 42 | 2
SGPT increased (Metabolism and nutrition disorders) | 47 | 4
Weight loss (Metabolism and nutrition disorders) | 29 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 91 | 55
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 12
Anxiety (Nervous system disorders) | 28 | 5
Depression (Nervous system disorders) | 31 | 14
Dizziness (Nervous system disorders) | 37 | 16
Insomnia (Nervous system disorders) | 39 | 16
Cough increased (Respiratory, thoracic and mediastinal disorders) | 100 | 40
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 54 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 52 | 4
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 53 | 18
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 48 | 18
Acne (Skin and subcutaneous tissue disorders) | 93 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 5
Rash (Skin and subcutaneous tissue disorders) | 73 | 14
Skin disorder (Skin and subcutaneous tissue disorders) | 26 | 18
Albuminuria (Renal and urinary disorders) | 166 | 45
Amenorrhea (Renal and urinary disorders) | 15/168 | 1/81
Dysuria (Renal and urinary disorders) | 30 | 10
Hematuria (Renal and urinary disorders) | 33 | 11
Impotence (Renal and urinary disorders) | 24/383 | 7/192
Kidney function abnormal (Renal and urinary disorders) | 73 | 47
Menorrhagia (Renal and urinary disorders) | 12/168 | 2/81
Metrorrhagia (Renal and urinary disorders) | 12/168 | 5/81
Ovarian cyst (Reproductive system and breast disorders) | 14/168 | 4/81
Local reaction to procedure (Injury, poisoning and procedural complications) | 42 | 25
Cellulitis (General disorders) | 31 | 6
Flu Syndrome (General disorders) | 62 | 30
Infection (General disorders) | 177 | 71
Sepsis (General disorders) | 28 | 6
Gastroenteritis (Gastrointestinal disorders) | 68 | 22
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 51 | 17
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 75 | 27
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 88 | 17
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 49 | 25
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 105 | 49
Fungal Dermatitis (Skin and subcutaneous tissue disorders) | 48 | 16
Herpes Simplex (Skin and subcutaneous tissue disorders) | 61 | 14
Herpes Zoster (Skin and subcutaneous tissue disorders) | 20 | 15
Urinary Tract Infection (Renal and urinary disorders) | 127 | 58
Skin Carcinoma (Skin and subcutaneous tissue disorders) | 18 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.